CLINICAL TRIAL: NCT00154843
Title: A Clinical Study to Determine Factors Affecting Absorption and Serum Levels of Lycopene After Supplementation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Urology, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 920704
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-01-14 (Estimated); Status verified 2006-08

CONDITIONS: BPH
Keywords: Lycopene; BPH; PSA; IPSS
MeSH Terms: interventions — Lycopene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Lycopene 15 mg/day
  Interventions: Drug: Lycopene
- B (Experimental): Lycopene 30 mg/day
  Interventions: Drug: Lycopene

INTERVENTIONS:
Drug: Lycopene — A: Lycopene15 mg/day ; B: Lycopene30 mg/day

SUMMARY:
Primary: To determine factors that affect absorption and serum levels of lycopene after supplementation.

Secondary:

1. To evaluate general safety and tolerability of oral lycopene 15 or 30 mg per day for 12 weeks.
2. To determine lycopene effects on reducing serum levels of prostate specific antigen (PSA) and on relieving lower urinary tract symptoms (LUTS) in relation to prostate hypertrophy as evaluated by the International Prostate Symptom Score (I-PSS).

DETAILED DESCRIPTION:
This is an uncontrolled intervention study in which eligible male subjects (N=60), after a two-week washout, will be randomized to receive lycopene either 15 or 30 mg per day for 12 weeks. About equal numbers of subjects will be randomized to either 15 or 30 mg of lycopene (about 30 subjects for each arm). The study is expected to be finished in 2 year. The study is expected to be finished in 2 year. Concerning an expected dropout rate of 10%, 66 subjects will be recruited for the study.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged 40 or older with no pathologically-proven prostate cancer or other cancers. Patients who have had a negative prostate biopsy are still acceptable.
* Subjects with a PSA between 2.5 and 20.0 ng/ml.
* Subjects understand the study procedures and agree to participate in the study by providing a written informed consent and scheduled blood or urine samples.
* Subjects whose liver function and renal function tests are within normal range.

Exclusion Criteria:

* Subjects who may have fluctuated serum PSAs, such as urinary tract infection, prostatitis, acute urinary retention, receiving radiotherapy to the pelvis, etc.
* Subjects who have received a prostate surgery or biopsy within 6 weeks before the initiation of lycopene supplementation.
* Subjects who may or will receive a prostate surgery or biopsy within 12 weeks of the initiation of lycopene supplementation.
* Subjects who have known allergic reaction to carotenoids including lycopene.
* Subjects who are participating or will participate in other clinical trials.
* Subjects who are taking medications that may alter serum PSA levels, such as 5-alpha reductase inhibitor (eg. finasteride), sex steroids or hormonal agents (eg. luteinizing hormone releasing hormone agonists, cyproterone acetate, flutamide, bicalutamide, megesterol acetate, etc.).
* Subjects who may require increased dosage of medications for lower urinary tract symptoms (LUTS) during the 12 weeks of protocol treatment. Subjects who have been put on medications for LUTS before entry and have a stabilized disease are still acceptable. These medications include, but note limited to, selective or non-selective alpha-blockers and anti-cholinergics.
* Subjects who have or have had clinical gastrointestinal malabsorption regardless of the etiology.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2004-03; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
serum lycopene levels | two years

SECONDARY OUTCOMES:
I-PSS, peak flow rate | two years

CONTACTS AND LOCATIONS:
Overall Officials: Yeong-Shiau Pu, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan